CLINICAL TRIAL: NCT06127446
Title: The Registry of Genetic Alterations of Taiwan Ovarian Cancer
Status: Recruiting | Type: Observational
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: National Taiwan University Hospital (Other); Mackay Memorial Hospital (Other); Cathay General Hospital (Other); China Medical University Hospital (Other); Taichung Veterans General Hospital (Other); National Cheng-Kung University Hospital (Other); Chang Gung Medical Foundation (Other); Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Sponsor
Other Study IDs: T1E23
Record Dates: First submitted 2023-10-25; First posted 2023-11-13 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-04

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer; Next generation sequencing
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Next-generation sequencing
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Despite recent progress in chemotherapy and targeted therapy for ovarian cancer, the 5-year survival rate remains around 40% because of rapid development of treatment resistance and recurrence. The sensitivity to platinum agents or BRCA genes mutation has been the prerequisite for improved survival using PARP inhibitors, though only 15-20% ovarian cancer patients harbor BRCA mutations through germline or somatic variants. Bevacizumab can only delayed disease recurrence but failed to improve overall survival. Several approved cancer therapeutics with established safety and toxicity profiles should be assessed in the immediate future based on biomarkers of platinum resistant, BRCA wild type recurrent ovarian cancer.

Furthermore, the proportion high grade serous and clear cell adenocarcinoma of ovary cancer in Taiwan increased substantially in recent 10 years. Genetic factors (such as homologous recombination deficiency, mismatch repair genes mutation), environmental factors (such as oral contraceptives, nulliparity/low parity) as well as comorbidity including endometriosis may be associated with the changing pattern and clinical outcomes of ovarian cancer in Taiwan.

Next-generation sequencing technology has enabled cancer genome sequencing in screening and searching for new cancer genes in an efficient manner. This massive sequencing technique not only help to identify new altered genes for novel biomarker development, but also reveal gene alterations sensitive or resistant to specific therapies.

The specific aims of this project are (1) to systemically explore genomic profiling of Taiwanese primary or platinum-resistant or -sensitive recurrent (or recurrent) ovarian cancer focusing on high grade serous and clear cell adenocarcinoma; (2) to collect clinical data regarding comorbidity, survival time and responses to major types of anticancer therapy; and (3) to establish a comprehensive ovarian cancer cohort for additional translational studies. The long-term goals of this study are to help implement personalized therapy, to develop novel therapy, and to improve outcomes of patients with ovarian cancer.

DETAILED DESCRIPTION:
Development of an integrated database of genetic background from treatment-naïve or recurrent populations, clinical information, and therapeutic outcomes in primary and recurrent ovarian cancer of high grade serous or clear cell adenocarcinoma.

1. To enroll 300 patients who fit the criteria of this study in the enrolled period.
2. To perform large-scale NGS analysis including 440 cancer gene panel and 24 HRD panel for specific populations, to create a map containing important genetic characteristics to help understand the mechanisms of drug resistance, and to find novel treatment strategies.
3. To collect tumor, non-tumor normal tissues and/or blood sample for genetic study (including NGS, whole-exome sequencing, RNA sequencing), proteomic study (including phosphoprotein), human leukocyte antigen testing, neoantigen and biomarker analyses.
4. To record previous therapeutic agents and accompanying treatment response and adverse events

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and above.
2. Stage I to IV high grade serous or clear cell carcinoma of ovary, peritoneal and fallopian tube.
3. Patients with primary ovarian cancer had undergone primary surgery. Patients with recurrent ovarian cancer had undergone primary surgery (and biopsy/surgery for recurrent tumors).
4. Tumor tissues before neoadjuvant therapy will be collected for patients receiving surgery after any neoadjuvant treatment.
5. Willingness to provide the surgical tissues of primary tumors, non-tumor part normal tissue (and paired recurrent tumors in 80 patients).
6. Willingness to provide blood sample of 20ml within four weeks after registration (in at least 72 patients of primary ovarian cancer and 72 patients of recurrent ovarian cancer).
7. Patient fully understand the protocol with the willingness to have regular follow-up.
8. Life expectancy more than 3 months.

Exclusion Criteria:

1. Concomitant ovarian and endometrial cancer
2. Paraffin tissue tumor block older than five years.
3. Tumor specimen of primary surgery or recurrent biopsy/surgery are not qualified for genetic testing.
4. Concomitant malignancy under surveillance or treatment in the past three years (excluding curatively treated basal or squamous cell skin carcinoma or carcinoma in situ)
5. Inability to cooperate or undesirable compliance to the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Ovarian cancer
Study Population: Stage I to IV high grade serous or clear cell ovarian cancer
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-12-13 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Large-scale NGS analysis for specific populations | 2023/10~2028/12
  Development of an integrated database of genetic background from treatment-naïve or platinum-refractory populations, clinical information, and therapeutic outcomes in primary and recurrent ovarian cancer of high grade serous or clear cell adenocarcinoma.

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Ju Ch'ang, Principal Investigator — National Health Research Institutes, Taiwan
Locations (8):
- Taiwan (8):
  - Chang Gung Medical Foundation, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Cathay General Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - National Taiwan University Hospital, Taipei